CLINICAL TRIAL: NCT04328662
Title: A National, Prospective, Non-interventional Study of NINLARO in Real World Clinical Practice
Brief Title: A Study of Ninlaro in Real World Clinical Practice in China
Status: Active, not recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: C16050; U1111-1237-5126 (Registry Identifier: WHO); EUPAS30733 (Registry Identifier: ENCEPP)
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma; Neoplasms, Plasma Cell
Keywords: Drug Therapy
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Participants with RRMM: Participants diagnosed with relapsed or refractory multiple myeloma (RRMM) who have received at least one dose of ixazomib plus lenalidomide - low dose dexamethasone (IRd) treatment, will be observed prospectively. Data will be collected from study sites such as clinical departments and pharmacies in hospitals as a part of routine clinical visits of participants to evaluate effectiveness and safety information.
- Cohort 2: Participants with NDMM, RRMM, and Non-myeloma: Participants diagnosed with NDMM who have received at least one dose of ixazomib-based regimen treatment, diagnosed with RRMM who have received at least one dose non-IRd ixazomib-based regimens treatment, and diagnosed with non-myeloma who have received at least one dose of ixazomib-based regimens treatment, will be observed prospectively. Data will be collected from study sites such as clinical departments and pharmacies in hospitals as a part of routine clinical visits of participants to evaluate effectiveness and safety information.

SUMMARY:
The main purpose of this study is to collect additional safety information of ixazomib citrate (Ninlaro) when used to treat multiple myeloma in real world clinical practice in China. Participants will be treated with Ninlaro according to the normal clinical practice during this study.

DETAILED DESCRIPTION:
This is a prospective, non-interventional study in Chinese participants with relapsed refractory multiple myeloma (RRMM), newly diagnosed multiple myeloma (NDMM) and non-myeloma who are undergoing or will receive at least one dose of ixazomib citrate. Data will be collected to assess safety information when NINLARO is used in the real world, based on known risks and missing safety information.

The study will enroll approximately 3000 patients. The data will be collected prospectively as part of routine clinical visits of participants. Participants will be assigned to one of the two observational cohorts:

* Cohort 1: Participants with RRMM
* Cohort 2: Participants with NDMM, RRMM, and Non-myeloma

The multi-center trial will be conducted in China. The overall duration of study will be approximately 64 months. All participants will be followed up for 21 months unless withdrawal of Informed Consent Form, loss of follow-up or death, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing treatment with Ninlaro (of less than 3 months from initial treatment with Ninlaro) or to be prescribed with Ninlaro capsule.
2. Participants will be able to sign Informed Consent Form to participate.

Exclusion Criteria:

1. Currently participates or plans to participate in any interventional clinical trial.
2. Any other reason that, in the Investigator's opinion, makes the participant unsuitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese participants with RRMM who have received at least one dose of IRd or non-IRd ixazomib based regimen treatment, and NDMM and non-myeloma who have received at least one dose of ixazomib-based regimen treatment will be observed prospectively.
Sampling Method: Non-Probability Sample
Enrollment: 482 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who Have one or More Adverse Events | From signing of the informed consent to 60 days after administration of the last dose of NINLARO (Up to Month 64)

SECONDARY OUTCOMES:
Number of Participants Reporting one or More Serious Adverse Events (SAEs), Adverse Drug Reaction (ADRs) and Adverse Events of Special Interest (AESI) | From signing of the informed consent to 60 days after administration of the last dose of NINLARO (Up to Month 64)
Number of Participants With Dose Adjustments During the Study | Up to Month 64
Number of Participants Categorized by Clinical Characteristics | Up to Month 64
Number of Participants Based on Disease Characteristics | Up to Month 64
Number of Participants With Multiple Myeloma Treatment | Up to Month 64
Overall Survival (OS) | From the date of sign Informed Consent Form to the date of death due to any cause (Up to Month 64)
  OS is measured as the time from the date of sign Informed Consent Form to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (28):
- China (28):
  - Anhui Cancer Hospital, Hefei, Anhui
  - Beijing Chao-yang Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Jishuitan Hospital, Beijing, Beijing Municipality
  - Beijing Chao-yang Hospital,Capital Medical University(Shijingshan), Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Sun Yat-Sen Memorial Hospital, Guangzhou, Guangdong
  - Zhujiang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Hainan General Hospital, Haikou, Hainan
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Soochow Hongci Blood Disease Hospital, Suzhou, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Affiliated Hospital of Jining Medical College, Jining, Shandong
  - Tai'an Central Hospital, Tai’an, Shandong
  - Zhabei Central Hospital, Jing'an District, Shanghai, Shanghai, Shanghai Municipality
  - Datong Third People's Hospital, Datong, Shanxi
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Shaoxing People's Hospital, Shaoxing, Zhejiang
  - Taizhou First People's Hospital, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/